CLINICAL TRIAL: NCT05649748
Title: An Open-Label Extension Study to Assess the Safety, Tolerability, and Effectiveness of the Long-Term Use of Treprostinil Palmitil Inhalation Powder in Participants With Pulmonary Arterial Hypertension
Brief Title: An Extension Study of Treprostinil Palmitil Inhalation Powder (TPIP) for Pulmonary Arterial Hypertension (PAH)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS1009-203; 2022-001951-18 (EudraCT Number); 2023-505539-11-00 (Other: EU CT Number)
Expanded Access: NCT06939647 (Available)
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Treprostinil Palmitil
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treprostinil Palmitil Inhalation Powder (TPIP) (Experimental): Participants who are not transitioning immediately from other TPIP studies:INS1009-201(NCT04791514), INS1009-202(NCT05147805) and other lead-in studies, will be given TPIP, once daily (QD), starting with 80 micrograms (μg), up-titrated to highest tolerated dose between 80 μg and 640 μg during 3-week titration period that maybe increased upto maximum dose of 1280 μg QD post initial titration, per investigator's assessment. Overall treatment period=24 months.
  Participants transitioning immediately from randomized blinded lead-in TPIP study and who previously received:
  1. TPIP- will be given placebo QD(80 μg upto achieved TPIP dose from previous study)along with achieved TPIP dose from previous study in blinded manner during 3-week titration period.
  2. Placebo- will be given TPIP QD (80 μg up to achieved placebo dose from previous study)along with achieved placebo dose from previous study in blinded manner during 3-week titration period.Overall treatment period=24 months.
  Interventions: Drug: Treprostinil Palmitil; Drug: Placebo

INTERVENTIONS:
Drug: Treprostinil Palmitil — Administered by oral inhalation, using a Plastiape capsule-based dry powder inhaler.
  Other Names: INS1009
Drug: Placebo — Administered by oral inhalation using a Plastiape capsule-based dry powder inhaler

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of the long-term use of TPIP in participants with PAH from studies INS1009-201 (NCT04791514), INS1009-202 (NCT05147805) and other lead-in studies of TPIP in participants with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who completed end of treatment study visit in Study INS1009-201, INS1009-202, or any other lead-in PAH TPIP study. Participants for whom the OLE study was not available at the time of their completion of the lead-in study are eligible for enrolment within one year of their lead-in end of treatment visit.
* Complete baseline screening assessments to confirm eligibility to participate if more than 30 days have elapsed since the end of the study visit in Study INS1009-201, INS1009-202, or any other lead-in PAH TPIP study.

Exclusion Criteria:

* Initiation of parenteral administration of prostacyclin analogues (eg, TRE, epoprostenol) since the completion of studies INS1009-201, INS1009-202 or other TPIP studies. Initiation of inhaled prostacyclin analogues (eg, TRE [Tyvaso] or iloprost) and oral prostacyclin analogues (eg, TRE [Orenitram]) or receptor agonists (eg, selexipag) are permitted if stopped 24 hours prior to the start of study drug administration.
* Any new ventricular or supraventricular tachyarrhythmia except for paroxysmal atrial fibrillation and any new symptomatic bradycardia.
* New-onset of heart disease including left ventricular ejection fraction (LVEF) ≤40% or clinically significant valvular, constrictive, or symptomatic atherosclerotic heart disease (eg, stable angina, myocardial infarction, etc).
* New evidence of thromboembolic disease as assessed by ventilation/perfusion (VQ) scan, pulmonary angiography, or pulmonary computed tomography (CT) scan.
* Active and current symptomatic coronavirus disease 2019 (COVID-19) or previous severe disease and/or hospitalization due to COVID-19.
* Interval organ transplantation.
* New active liver disease or hepatic dysfunction.
* Interval malignancy with exception of completely treated in situ carcinoma of the cervix and completely treated non-metastatic squamous or basal cell carcinoma of the skin.
* Use of any investigational drug/device or participation in any investigational study within 30 days prior to screening, not including TPIP of the lead-in study.
* Current use of cigarettes (as defined by Centers for Disease Control and Prevention [CDC]) or e-cigarettes: An adult who has smoked at least 100 cigarettes in his or her lifetime, who smokes either every day or some days.
* Participants who currently inhale marijuana (recreational or medical).

Note: Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience at Least one Treatment Emergent Adverse Event (TEAE) and TEAEs by Severity | From screening up to last follow up visit (Up to approximately 26 months)

SECONDARY OUTCOMES:
Absolute Change From Pre-Open Label Extension (OLE) Baseline in 6-Minute Walk Distance (6MWD) | Pre-OLE baseline (baseline of the lead-in TPIP study), Months 6, 12, 18, and 24
Relative Change From Pre-OLE Baseline in 6MWD | Pre-OLE baseline (baseline of the lead-in TPIP study), Months 6, 12, 18, and 24
Change From Pre-OLE Baseline in the Concentration of N-Terminal Fragment B-Type Natriuretic Peptide (NT-proBNP) in Blood | Pre-OLE baseline (baseline of the lead-in TPIP study), Months 6, 12, 18, and 24
Change From Pre-OLE Baseline in the Registry to Evaluate Early and Long-Term PAH Disease Management (REVEAL) Lite 2.0 Score | Pre-OLE baseline (baseline of the lead-in TPIP study), Months 6, 12, 18, and 24
Change From Pre-OLE Baseline in New York Heart Association/ World Health Organization (NYHA/WHO) Functional Capacity Class | Pre-OLE baseline (baseline of the lead-in TPIP study), Months 6, 12, 18, and 24
Annualized Clinical Worsening Event Rate | OLE Baseline (Day 1) up to Month 24 or early discontinuation
  Annualized clinical worsening event rate is defined as the total number of clinical worsening events that occurred during the treatment period divided by the total number of participant-years during the treatment period. Clinical worsening events are one of the following: All-cause death, or onset of TEAE with a fatal outcome occurring ≤ 14 days after study drug discontinuation; Hospitalization for right heart failure (for > 48 hours), heart-lung or lung transplant, or atrial septostomy; Addition (or increase in dose) of specified PAH-specific medications; Combined occurrence of events including ≥20% decrease in 6MWD, worsening WHO/NYHA functional capacity class, and appearance of or worsening of signs/symptoms of right heart failure from baseline.
Plasma Concentration Levels of Treprostinil Palmitil (TP) and Treprostinil (TRE) | OLE Baseline (Day 1), Months 6, 12, 18, and 24

CONTACTS AND LOCATIONS:
Locations (45):
- United States (6):
  - USA005, Jacksonville, Florida
  - USA011, Tampa, Florida
  - USA006, Chicago, Illinois
  - USA001, Chicago, Illinois
  - USA102, New York, New York
  - USA016, Dallas, Texas
- Argentina (5):
  - ARG009, Quilmes, Buenos Aires
  - ARG006, Rosario, Santa Fe Province
  - ARG007, San Miguel de Tucumán, Tucumán Province
  - ARG004, Córdoba
  - ARG001, Córdoba
- Austria (2):
  - AUT002, Linz, Upper Austria
  - AUT001, Vienna
- BEL003, Brussels, Belgium
- Brazil (3):
  - BRA004, Belo Horizonte, Minas Gerais
  - BRA006, Porto Alegre, Rio Grande do Sul
  - BRA002, Blumenau, Santa Catarina
- DNK001, Aarhus, Central Jutland, Denmark
- Germany (3):
  - GER005, Heidelberg, Baden-Wurttemberg
  - GER003, München, Bavaria
  - GER002, Lübeck, Schleswig-Holstein
- Italy (4):
  - ITA002, Pavia, Lombardy
  - ITA005, Monza
  - ITA001, Palermo
  - ITA004, Roma
- Japan (6):
  - JPN005, Sapporo, Hokkaido
  - JPN004, Sapporo, Hokkaido
  - JPN007, Kurume-shi, Hukuoka
  - JPN006, Tsukuba, Ibaraki
  - JPN002, Okayama, Okayama-ken
  - JPN003, Suita-Shi, Osaka
- Malaysia (3):
  - MYS005, Alor Star, Kedah
  - MYS002, Kuantan, Pahang
  - MYS004, Sungai Buloh, Selangor
- Mexico (4):
  - MEX005, Lomas de Guevara, Jalisco
  - MEX001, Monterrey, Nuevo León
  - MEX003, Mexico City
  - MEX004, San Luis Potosí City
- Philippines (2):
  - PHL001, Quezon City, National Capital Region
  - PHL002, Makati City
- Serbia (2):
  - SRB001, Belgrade
  - SRB003, Belgrade
- Spain (2):
  - ESP001, Santander
  - ESP003, Seville
- GBR001, Bath, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: No